CLINICAL TRIAL: NCT02967536
Title: Investigating the Neuropathology of Obstructive Sleep Apnoea
Acronym: INcOSA
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 170912
Record Dates: First submitted 2016-08-17; First posted 2016-11-18 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Obstructive Sleep Apnoea; Inflammation
Keywords: cognitive function; microglia; neuroinflammation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participants will be invited to donate samples (blood or saliva) to the Biomedical Research Centre (BRC) Bioresource. In order to have statistical power for genetic analysis, samples from INcOSA participants will need to be combined with those from the OSA BioResource (Research Tissue Bank) volunteers who have provided consented biological samples for future research.
  These samples may be used for genetic, epigenetic, metabolomic or proteomic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mild OSA: Untreated OSA patients. Apnoea-Hypopnoea Index (AHI) >5 events/hour and <10 events/hour with Epworth Sleepiness Score (ESS)>9.
- Severe OSA: Untreated OSA patients. AHI >30 events/hour, with excessive sleepiness (ESS >9).
- Healthy control: Healthy control. AHI <5 events/hour.

SUMMARY:
Our multi-disciplinary research group works closely with people who have obstructive sleep apnoea. This is a life-long illness that causes breathing to stop during sleep, which leads to low-oxygen in the blood. Breathing restarts when the airway at the back of the throat reopens, usually during arousal from sleep. In some people the repeated arousals from sleep cause daytime sleepiness. Our research has shown that the low blood oxygen levels affect thinking and feeling, and in some cases we think it damages the brain cells involved with memory, attention, emotions and decision-making.

This study will investigate the relationship between the amount of oxygen in the blood and the loss (if any) of brain cells. Also how the ability to perform complex tasks is affected in patients that suffer from sleep apnoea. The results will show whether the brain damage in patients with sleep apnoea can be reversed with treatment. These findings will guide doctors in the treatment for sleep apnoea and they will cast light onto the process of memory decline with the aim to preserve brain function.

DETAILED DESCRIPTION:
This is a cross-sectional physiological study, which is anticipated to last for 4 years. In order to study the mechanism of cognitive dysfunction in Obstructive Sleep Apnoea (OSA), patients will start Continuous Positive Airway Pressure (CPAP) treatment following the confirmed diagnosis of sleep apnoea. CPAP is the treatment of choice for patients with moderate to severe OSA who are sleepy during the day. It is also used in patients with mild OSA if they are excessively sleepy or suffer from cardiovascular risk factors. It is recommended by the National Institute for Clinical Excellence (NICE) as a treatment for adults with moderate or severe OSA (Sleep apnoea - continuous positive airway pressure, NICE 2008). In the proposed study the initiation of CPAP will be within the 18 week period set out in the National Health Service (NHS) Improvement Plan and Standards for Better Health (Standards for Better Health, Department of Health 2004). No patient with a diagnosis of OSA will commence treatment with CPAP later than advised by the NICE guidelines of clinical judgement for the best interest of the patient.

In order to investigate the neuroinflammation process and discrete changes in the brain of patients with OSA, a minimum of 9 patients with mild OSA and 9 patients with severe OSA will be compared to 9 healthy controls following initial sleep (assessment) study. All participants will undergo a dynamic Positron Emission Tomography with Magnetic Resonance Imaging (PET-MR) scan with the Translocator protein (TSPO) tracer [Fluorine-18] N,N-diethyl-2-[4-(2-fluoroethoxy)phenyl]-5,7-dimethylpyrazolo[1,5-a]pyrimidine-3-acetamide (DPA-714) at the time of enrolment to the study. Each participant will also have an MRI scan and cognitive testing.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants with OSA:

* Male patients
* With untreated OSA either mild (AHI≥5/hour and ≤10/hour)
* or severe (AHI≥30/hour)
* With excessive sleepiness (ESS≥9)
* Aged 18-69 years

Healthy control group:

* Male participants
* No history of sleep disorders
* AHI≤5/hour
* No current or previous major neurological or psychiatric disease
* Not currently undertaking neuropharmacological treatment
* Non-smoker
* No history of alcohol or recreational drug abuse
* No major organ failure
* Not professional drivers or shift workers

EXCLUSION CRITERIA:

* Having other sleep disorders, neurological or psychiatric disease
* Undertaking neuropharmacological treatment
* Has a history of alcohol or recreational drug abuse, major organ failure
* Professional drivers or shift workers
* Unable to have MR scan (e.g. too heavy (>200Kg) or have ferromagnetic implants)
* [18F]DPA-714 affinity too low
* Inability to comprehend what is proposed
* Inability to travel to the research sites

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient group:
  * Untreated patients with mild Sleep Apnoea - Apnoea-Hypopnoea Index (AHI) >5 events/hour and <10 events/hour with excessive sleepiness (Epworth sleepiness score >9).
  * Untreated patients with severe Sleep Apnoea - AHI >30 events/hour with excessive sleepiness (Epworth sleepiness score >9).
  Healthy control group:
  * Male participants
  * No history of sleep disorders
  * AHI≤5/hour
  * No current or previous major neurological or psychiatric disease
  * Not currently undertaking neuropharmacological treatment
  * Non-smoker
  * No history of alcohol or recreational drug abuse, major organ failure
  * Not professional drivers or shift workers.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Levels of neuroinflammation, brain morphology and neurophysiology will be measured via MRI, PET-MRI imaging & EEG. | MRI, PET-MRI & EEG data analyses will begin right after the completion of data collection, and the summary of results will be reported as soon as available, expected before the completion date of the study as per IRAS 01/06/2020.
  27 participants, 9 healthy controls, 9 mild patients & 9 severe patients.
Cognitive performance using the CANTAB battery. | Cognitive performance data analyses will be conducted after the completion of data collection, and the summary of results will be reported along the rest of results in the summary that will be published before 01/06/2020.
  27 participants, 9 healthy controls, 9 mild patients & 9 severe patients.

SECONDARY OUTCOMES:
Genetic analysis and linkage to clinical and neuroimaging data will be measured using biological samples (blood or saliva) analysed and stored in the BioResource for Mental and Neurological Health. | Genetic analysis and linkage to clinical and neuroimaging data analyses are expected to continue after the end of the primary study and they will be independently reported by the BioResource for Mental and Neurological Health KCL, within 5 years of study
  18 patients, 9 mild & 9 severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Rosenzweig, MD, PhD, Principal Investigator — King's College London
Locations (1):
- Guy's Hospital Sleep Centre, London, United Kingdom